CLINICAL TRIAL: NCT03635619
Title: 3 T MRI in the Preoperative TN Staging and Prediction of Response to Neoadjuvant Therapy in Patients With Esophageal Cancer
Brief Title: The Application of 3T MRI in Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: FSK001
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2019-08

CONDITIONS: Esophageal Cancer TNM Staging; Magnetic Resonance Imaging; Prognosis
Keywords: Esophageal Cancer; Magnetic Resonance Imaging; Prognosis; neoplasm staging
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
It is very significant that assessing TN staging in esophageal cancer patients before surgery, furthermore, determining the optimize surgical strategy, predict the the efficacy of radiotherapy for patients who were not chosen to be surgeried, and define the range of lymph node for radiotherapy. It has been reported that the application of MRI in metastasis of lymph node of other cancer, but not in metastasis lymph node with esophageal cancer. Only a few studies focused on T staging using conventional MRI in esophageal cancer, however, relatively new sequences in the chest deserve widely used. To develop a pre-treatment evaluation methods for TN staging in patient with esophageal cancer by utilization of the new imaging methods (T2-TSE-BLADE, T2 maps, StarVIBE). By analysising the relationship between TN staging and imaging features to find the imaging characteristics for TN staging, and to find the indicators of magnetic resonance imaging new technology and reference values for facilitate pre-treatment diagnosis of lymphnode metastasis, optimize surgical strategy, predict the the efficacy of adjunctive therapy, and OS and define the range of lymph node for radiotherapy, as making personal treatment planning for esophageal cancer.

DETAILED DESCRIPTION:
To explore the value of 3 T MRI using multiple sequences, including T2-TSE-BLADE, T2 maps and StarVIBE, in evaluating the preoperative TN staging and prediction of response to neoadjuvant therapy and OS in patients with esophageal cancer.

Patients with endoscopically biopsy-proven EC were prospectively enrolled for imaging on a 3 T scanner. The MRI protocol included T2-TSE-BLADE, T2 maps and StarVIBE sequences, and so on. Patients received treatment according to NCCN guideline. Readers assigned a TN stage on MRI, and post-operative pathologic confirmation was considered the gold standard. Inter-reader agreement, the diagnostic accuracy of TN staging on MRI were analyzed and compared to post-operative pathologic TN staging. MRI features were analyzed to find the correlation between pretreatment MRI features and response or OS. The study will includ 400 patients. Inter-reader agreements of TN staging were analyzed excellent for MRI. Diagnostic accuracy of MRI will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients with preoperative pathologically con-firmed EC by endoscopy and preoperative imaging data (esophagography\CT\EUS\MRI) were included.
2. No contraindications for MRI examination.
3. The patients participate in this study with informed consent.

Exclusion Criteria:

1. The patients couldn't performed MR scanning or artefacts affect the evaluation.
2. ThePatients are extremely anxious and uncooperative about surgery or neoadjuvant therapy.
3. PatientsThe patients refuse to participate in the project.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with endoscopically biopsy-proven EC will receive treatment.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-09-02 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
MRI TN staging in Esophageal Cancer | Sep 1, 2018-Dec 31, 2019
  To explore the value of 3 T MRI using multiple sequences in evaluating the preoperative TN staging of esophageal cancer treated with surgery, with pathologic confirmation

SECONDARY OUTCOMES:
MRI prediction of prognosis in esophageal cancer | Sep 1, 2018-Dec 31, 2020
  To explore the value of 3 T MRI using multiple sequences in predicting the response and OS of esophageal cancer treated with surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Baoxia He, MD, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dumont P, Wihlm JM, Hentz JG, Roeslin N, Lion R, Morand G. Respiratory complications after surgical treatment of esophageal cancer. A study of 309 patients according to the type of resection. Eur J Cardiothorac Surg. 1995;9(10):539-43. doi: 10.1016/s1010-7940(05)80001-6. PMID 8562096
- [Background] Wu CC, Chen CJ. Esophageal carcinoma. N Engl J Med. 2015 Apr 9;372(15):1472. doi: 10.1056/NEJMc1500692. No abstract available. PMID 25853761
- [Background] Omloo JM, Lagarde SM, Hulscher JB, Reitsma JB, Fockens P, van Dekken H, Ten Kate FJ, Obertop H, Tilanus HW, van Lanschot JJ. Extended transthoracic resection compared with limited transhiatal resection for adenocarcinoma of the mid/distal esophagus: five-year survival of a randomized clinical trial. Ann Surg. 2007 Dec;246(6):992-1000; discussion 1000-1. doi: 10.1097/SLA.0b013e31815c4037. PMID 18043101
- [Background] Allum WH, Blazeby JM, Griffin SM, Cunningham D, Jankowski JA, Wong R; Association of Upper Gastrointestinal Surgeons of Great Britain and Ireland, the British Society of Gastroenterology and the British Association of Surgical Oncology. Guidelines for the management of oesophageal and gastric cancer. Gut. 2011 Nov;60(11):1449-72. doi: 10.1136/gut.2010.228254. Epub 2011 Jun 24. No abstract available. PMID 21705456
- [Background] Chen J, Chen C, Xia C, Huang Z, Zuo P, Stemmer A, Song B. Quantitative free-breathing dynamic contrast-enhanced MRI in hepatocellular carcinoma using gadoxetic acid: correlations with Ki67 proliferation status, histological grades, and microvascular density. Abdom Radiol (NY). 2018 Jun;43(6):1393-1403. doi: 10.1007/s00261-017-1320-3. PMID 28939963
- [Background] Cassinotto C, Feldis M, Vergniol J, Mouries A, Cochet H, Lapuyade B, Hocquelet A, Juanola E, Foucher J, Laurent F, De Ledinghen V. MR relaxometry in chronic liver diseases: Comparison of T1 mapping, T2 mapping, and diffusion-weighted imaging for assessing cirrhosis diagnosis and severity. Eur J Radiol. 2015 Aug;84(8):1459-1465. doi: 10.1016/j.ejrad.2015.05.019. Epub 2015 May 19. PMID 26032126
- [Background] Zhang H, Xue H, Alto S, Hui L, Kannengiesser S, Berthold K, Jin Z. Integrated Shimming Improves Lesion Detection in Whole-Body Diffusion-Weighted Examinations of Patients With Plasma Disorder at 3 T. Invest Radiol. 2016 May;51(5):297-305. doi: 10.1097/RLI.0000000000000238. PMID 26704452
- [Background] Li X, Qu JR, Luo JP, Li J, Zhang HK, Shao NN, Kwok K, Zhang SN, Li YL, Liu CC, Zee CS, Li HL. Effect of intravenous gadolinium-DTPA on diffusion-weighted imaging of brain tumors: a short temporal interval assessment. J Magn Reson Imaging. 2014 Sep;40(3):616-21. doi: 10.1002/jmri.24386. Epub 2013 Oct 31. PMID 24925118
- [Background] Zhang F, Qu J, Zhang H, Liu H, Qin J, Ding Z, Li Y, Ma J, Zhang Z, Wang Z, Zhang J, Zhang S, Dong Y, Grimm R, Kamel IR, Li H. Preoperative T Staging of Potentially Resectable Esophageal Cancer: A Comparison between Free-Breathing Radial VIBE and Breath-Hold Cartesian VIBE, with Histopathological Correlation. Transl Oncol. 2017 Jun;10(3):324-331. doi: 10.1016/j.tranon.2017.02.006. Epub 2017 Mar 19. PMID 28327459